CLINICAL TRIAL: NCT07220096
Title: Registry Trial and Needs Assessment of Patients With Young-onset Lung Cancer: Impact of a Dedicated Care Program on Patient Experience and Outcomes
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-0646; NCI-2025-07304 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-09-30; First posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Assessment of Patients with Young-Onset Lung Cancer: This is a registry trial enrolling participants with NSCLC diagnosed and histologically confirmed prior to the age of 50 years identified. Each participant will participate in an intake survey as well as periodic recurring surveys to provide feedback to the YOLC Program, to elucidate the individual participant's care needs, and to assess changes in personal goals, wellness, financial impact, and family support over time
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Participants will complete an intake survey and repeat surveys at the following time points:
  * Baseline
  * 3 months
  * 6 months
  * 9 months
  * 12 months
  * 18 months
  * 24 months
  * 36 months
  * 48 months
  * 60 months

SUMMARY:
The goal of this research study is to learn about:

The effect of enrolling in the YOLC program on patient satisfaction with care provided,

The needs of patients younger than 50 with lung cancer and their family, and

The impact of participating in peer support networks on these patients.

DETAILED DESCRIPTION:
Primary Objectives:

1. To determine whether enrollment in a dedicated program (YOLC) results in improved patient satisfaction with care provided.
2. To characterize the distinct needs of patients under age 50 diagnosed with lung cancer as well as those of their families, and how these needs may change over time throughout the care pathway.
3. To evaluate the impact of participation in peer support networks and whether it has a beneficial effect on the primary and secondary endpoints.

Secondary Objectives:

1. To determine whether enrollment in a dedicated program (YOLC) results in improved patient satisfaction with care provided.
2. To characterize the distinct needs of patients under age 50 diagnosed with lung cancer as well as those of their families, and how these needs may change over time throughout the care pathway.
3. To evaluate the impact of participation in peer support networks and whether it has a beneficial effect on the primary and secondary endpoints.
4. Overall survival, defined by time from diagnosis to death from any cause
5. Clinical trial enrollment, defined by participation in any therapeutic clinical trial related to lung cancer treatment after diagnosis
6. Completion of multi-disciplinary consultations, defined by patients completing consultations with at least one other specialist other than a thoracic medical oncologist or thoracic surgeon from time of initial consultation for the YOLC Program
7. Quality of life, as defined by FACT-LUNG
8. Financial toxicity, as defined by patient-reported financial burden, including out-of-pocket costs, insurance coverage issues, and impact of overall financial well-being (measured using validated financial toxicity scale such as COST-FACIT

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years and under 50 years
* Histologic confirmation of NSCLC
* Able to complete an English-language survey independently or with the assistance of a native-language interpreter
* Pregnant women- may be enrolled due to age range of subjects. (Low risk)

Exclusion Criteria:

* Medical, psychiatric, cognitive, or other conditions that compromise the patient's ability to understand the patient information, to give informed consent, to comply with the study protocol or to complete the study.
* The following special patient population will be excluded from study group:

  * Individuals who are not yet adults (infants, children, teenagers)
  * Prisoners
  * Cognitively-impaired adults

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: MD Anderson
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2031-05-31 (Estimated)

PRIMARY OUTCOMES:
Participant satisfaction with care | Through study completion; an average of 5 year
  Assessed via validated survey instruments (e.g., FACT-L, COST-FACIT).
  • Focus on detecting even small changes in survey responses over time (baseline, 3, 6, 9, 12 months, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Eric Singhi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org